CLINICAL TRIAL: NCT06032715
Title: Brief Intervention for Reducing Prolonged Use of Sleep Medication Among Elderly
Brief Title: Brief Intervention for Sleep Medication Misuse Among Elderly
Acronym: BI-sleep
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Christofer Lundqvist, Professor, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: BI-sleep
Record Dates: First submitted 2023-08-17; First posted 2023-09-13 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Harmful Use of Hypnotic
Keywords: Z-hypnotics; insomnia; sleep; side effects; cognitive function; pain; behavioral intervention; dependence; quality of life
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Pain | interventions — Crisis Intervention

STUDY DESIGN:
Intervention Model Description: Parallel masked and controlled first part intervention vs Business as usual with follow-up after 6 months by masked assessors. Subsequently open single cross-over of business as usual patients to also receive the same intervention.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: GPs will be cluster randomized based on GP to two sequential teaching programs to learn the Brief Intervention procedure. The patients of those who have the course first will constitute the intervention arm while patients of GPs who are in the second course will constitute parallel business as usual controls in the masked part of the study. When the second group of GPs have their course, open cross-over will be possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI (Brief Intervention) (Active Comparator): Patients whose GPs have been taught the behavioral BI intervention aiming to reduce prolonged use of Z-hypnotics.
  Interventions: Behavioral: BI (Brief Intervention)
- BAU (Business as usual) (No Intervention): Patients whose GPs have not yet been taught the BI intervention. Patients only assessed in parallel with BI group by masked assessors using same instruments as for active comparator.
  This group also constitutes an open cross-over group to active intervention once the masked 6 months phase is completed.

INTERVENTIONS:
Behavioral: BI (Brief Intervention) — Short structured individual behavioral intervention to reduce inappropriate usage of Z-hypnotics
  Arms: BI (Brief Intervention)

SUMMARY:
Randomized controlled trial to evaluate effectiveness of behavioral Brief Intervention administered by General practitioners (GPs) versus business as usual on use of Z-hypnotics by elderly patients in primary care.

DETAILED DESCRIPTION:
Two armed study with controlled masked first part over 6 months. Active arm is with Brief Intervention for inappropriate use of Z-hypnotics among elderly with intervention delivered by trained GPs. Control arm is for patients handled by their (non-trained) GPs with business as usual (BAU). Main outcome is 6 weeks after intervention with additional data collection points after 6 months (blinded) and long-term follow-up to 12 months (open). After 6 months there will be an open single crossover as BAU GPs will then also receive training in the Brief Intervention method.

Baseline assessments are limited to self reports and automatic sleep assessment with actigraphy to avoid assessment effects. Follow-up at main outcome time point is in person, some outcomes are also by telephone assessment and compared to baseline prior to intervention (e g Actigraphy assessment.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported use of Z-hypnotics > 4 days per week and > 4 weeks

Exclusion Criteria:

* diagnosis of dementia,
* diagnosis of psychosis,
* diagnosis of major depression,
* diagnosis of delirium,
* unable to give informed consent,
* insufficient Norwegian language capacity to complete tests

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Inappropriate Z-hypnotics use | 6 weeks
  Proportion of patients with prolonged use of Z-hypnotics

SECONDARY OUTCOMES:
Pain visual analogue scale (VAS) | 6 weeks
  VAS assessment of experienced pain (1-100 mm, no pain (0), worst possible pain (100))
Cognitive function | 6 weeks
  Cognistat test total score (0-84, 84 best)
Cognitive function | 6 months
  Cognistat test total score (0-84, 84 best)
Experience of sleep | 6 weeks
  Global Sleep Assessment Questionnaire score (GSAQ) (11 items, Never, sometimes, usually, always. Item responses were converted to a common 0-100 scale, with a higher score indicating greater likelihood for presence of the disorder. .)
Experience of sleep | 6 months
  Global Sleep Assessment Questionnaire score (GSAQ) (11 items, Never, sometimes, usually, always. Item responses were converted to a common 0-100 scale, with a higher score indicating greater likelihood for presence of the disorder. .)
Sleep efficiency (random subpopulation) | 6 weeks
  Actigraphy assessed before and after intervention
Change compared to baseline of Z-hypnotics use | 6 weeks
  Proportion of patients with prolonged use of Z-hypnotics
Change compared to baseline of Z-hypnotics use | 6 months
  Proportion of patients with prolonged use of Z-hypnotics
Inappropriate Z-hypnotics use | baseline
  Proportion of patients with prolonged use of Z-hypnotics

OTHER OUTCOMES:
Quality of life measure, index | 6 months
  Euro QoL, five dimension, 5 level version (EQ-5D-5L index, Norwegian population norms valuation), 0-1 with 1 representing perfect health
Quality of life measure, VAS | 6 months
  Euro QoL, five dimension, 5 level version (EQ-5D VAS), 0-100 with 100 representing best health
Dependence score | 6 weeks
  Severity of dependence score (SDS), 0-15, 15 highest severity
Dependence score | 6 months
  Severity of dependence score (SDS), 0-15, 15 highest severity
MoCa score | 6 weeks
  Telefon - Montreal Cognitive Assessment (T-MoCA) for remote assessments. (0-22 points, normal cognition ≥ 18 / 22)
Self assessed cognitive function | 6 weeks
  Norwegian cognitive function instrument (KFI) (0-13 points yes=1 point, maybe=0,5 point, no=0 point)
Verbal fluency | 6 weeks
  FAS score (60 seconds timecap, using a cut-off score of 14 points indicating executive function deficits)
Multimorbidity | 6 weeks
  Cumulative Illness Rating Scale-Geriatric (CIRS-G) 0-56, 56 worst
Multimorbidity | 12 months
  Cumulative Illness Rating Scale-Geriatric (CIRS-G) 0-56, 56 worst
Polypharmacy | 6 weeks
  Number of regularly used medications
Readiness to change behaviour | Baseline
  Readiness to change behavior visual analogue scale scale, 0-100, 100 most ready
Prevalence of inappropriate medication use in screened population | At screening before baseline
  Patient self report in screening questionnaire
Prevalence self-reported sleep difficulties | At screening before baseline
  Patient self report in screening questionnaire
Anxiety and depression symptoms | 6 weeks
  Hospital anxiety and depression scale (HADS), 0-42, 42 worst
Anxiety and depression symptoms | 6 months
  Hospital anxiety and depression scale (HADS), 0-42, 42 worst
Mortality | 12 months, 24 months
  Based on automatic registration in electronic patient journal
Cognitive function, subdimensions | 6 weeks
  Cognistat test, subdimensions score, higher score is better cognitive function
Cognitive function, subdimensions | 6 months
  Cognistat test, subdimensions score, higher score is better cognitive function
Inappropriate Z-hypnotics use | 6 months
  Proportion of patients with prolonged use of Z-hypnotics
Pain visual analogue scale (VAS) | 12 months
  VAS assessment of experienced pain (1-100 mm, no pain (0), worst possible pain (100))
Cognitive function | 12 months
  Cognistat test total score (0-84, 84 best)
Inappropriate Z-hypnotics use | 12 months
  Proportion of patients with prolonged use of Z-hypnotics
Change compared to baseline of Z-hypnotics use | 12 months
  Proportion of patients with prolonged use of Z-hypnotics
Quality of life measure, index | 12 months
  Euro QoL, five dimension, 5 level version (EQ-5D-5L index, Norwegian population norms valuation)
Quality of life measure, VAS | 12 months
  Euro QoL, 0 (worse) - 100(best)score (EQ-5D VAS)
Experience of sleep | 12 months
  Global Sleep Assessment Questionnaire score (GSAQ) (11 items, Never, sometimes, usually, always. Item responses were converted to a common 0-100 scale, with a higher score indicating greater likelihood for presence of the disorder. .)
Pain visual analogue scale (VAS) | 6 months
  VAS assessment of experienced pain (1-100 mm, no pain (0), worst possible pain (100))

CONTACTS AND LOCATIONS:
Overall Officials: Christofer Lundqvist, MD, PhD, Study Chair — Akershus University Hospital and University of Oslo
Locations (1):
- Akershus University Hospital, Lørenskog, Norway

REFERENCES:
- [Background] Kristoffersen ES, Straand J, Vetvik KG, Benth JS, Russell MB, Lundqvist C. Brief intervention for medication-overuse headache in primary care. The BIMOH study: a double-blind pragmatic cluster randomised parallel controlled trial. J Neurol Neurosurg Psychiatry. 2015 May;86(5):505-12. doi: 10.1136/jnnp-2014-308548. Epub 2014 Aug 11. PMID 25112307
- [Background] Frich JC, Kristoffersen ES, Lundqvist C. GPs' experiences with brief intervention for medication-overuse headache: a qualitative study in general practice. Br J Gen Pract. 2014 Sep;64(626):e525-31. doi: 10.3399/bjgp14X681313. PMID 25179065
- [Background] Kristoffersen ES, Straand J, Vetvik KG, Benth JS, Russell MB, Lundqvist C. Brief intervention by general practitioners for medication-overuse headache, follow-up after 6 months: a pragmatic cluster-randomised controlled trial. J Neurol. 2016 Feb;263(2):344-353. doi: 10.1007/s00415-015-7975-1. Epub 2015 Dec 8. PMID 26645391
- [Background] Kristoffersen ES, Straand J, Russell MB, Lundqvist C. Lasting improvement of medication-overuse headache after brief intervention - a long-term follow-up in primary care. Eur J Neurol. 2017 Jul;24(7):883-891. doi: 10.1111/ene.13318. Epub 2017 May 23. PMID 28544265
- [Background] Cheng S, Siddiqui TG, Gossop M, Kristoffersen ES, Lundqvist C. The Severity of Dependence Scale detects medication misuse and dependence among hospitalized older patients. BMC Geriatr. 2019 Jun 24;19(1):174. doi: 10.1186/s12877-019-1182-3. PMID 31234786
- [Background] Siddiqui TG, Cheng S, Gossop M, Kristoffersen ES, Grambaite R, Lundqvist C. Association between prescribed central nervous system depressant drugs, comorbidity and cognition among hospitalised older patients: a cross-sectional study. BMJ Open. 2020 Jul 27;10(7):e038432. doi: 10.1136/bmjopen-2020-038432. PMID 32718926
- [Background] Siddiqui TG, Cheng S, Mellingsaeter M, Grambaite R, Gulbrandsen P, Lundqvist C, Gerwing J. "What should I do when I get home?" treatment plan discussion at discharge between specialist physicians and older in-patients: mixed method study. BMC Health Serv Res. 2020 Nov 3;20(1):1002. doi: 10.1186/s12913-020-05860-9. PMID 33143713
- [Background] Bjelkaroy MT, Cheng S, Siddiqui TG, Benth JS, Grambaite R, Kristoffersen ES, Lundqvist C. The association between pain and central nervous system depressing medication among hospitalised Norwegian older adults. Scand J Pain. 2021 Dec 16;22(3):483-493. doi: 10.1515/sjpain-2021-0120. Print 2022 Jul 26. PMID 34913326
- [Background] Siddiqui TG, Bjelkaroy MT, Cheng S, Kristoffersen ES, Grambaite R, Lundqvist C. The effect of cognitive function and central nervous system depressant use on mortality-A prospective observational study of previously hospitalised older patients. PLoS One. 2022 Mar 3;17(3):e0263024. doi: 10.1371/journal.pone.0263024. eCollection 2022. PMID 35239678
- See also: Humeniuk et al (2010), WHO: The Alcohol, Smoking and Substance involvement Screening Test (ASSIST): manual for use in primary care — https://apps.who.int/iris/handle/10665/44320
- See also: Babor et al (2001), WHO: Brief intervention for hazardous and harmful drinking : a manual for use in primary care — https://apps.who.int/iris/handle/10665/67210

DOCUMENTS (2):
  • Statistical Analysis Plan: Statistical analysis plan screening data (2024-08-23): https://cdn.clinicaltrials.gov/large-docs/15/NCT06032715/SAP_000.pdf
  • Statistical Analysis Plan: Statistical analysis plan main RCT (2024-11-13): https://cdn.clinicaltrials.gov/large-docs/15/NCT06032715/SAP_001.pdf